CLINICAL TRIAL: NCT06566222
Title: Chemoradiotherapy After Surgery Versus Preoperative Chemoradiotherapy for Stage II/III Mid-low Rectal Cancer With or Without High-risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChanghaiH-Radiotherapy
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NAT+High
  Interventions: Other: High-risk Factors
- NAT+Low
- PAT+High
  Interventions: Procedure: chemoradiotherapy after surgery; Other: High-risk Factors
- PAT+Low

INTERVENTIONS:
Procedure: chemoradiotherapy after surgery — chemoradiotherapy after surgery vs preoperative chemoradiotherapy
  Other Names: preoperative chemoradiotherapy
  Groups: PAT+High
Other: High-risk Factors — High-risk Factors vs low-risk Factors
  Other Names: low-risk Factors
  Groups: NAT+High; PAT+High

SUMMARY:
The purpose of this observational study is to understand the effect of different timing of chemoradiotherapy on overall survival in patients with stage II/III low- and medium-level rectal cancer with or without high-risk factors

ELIGIBILITY:
Inclusion Criteria:

1. The patient is between 18 and 80 years old;
2. Adenocarcinoma confirmed by pathology;
3. Colonoscopy or imaging examination confirmed that the distance between the lower edge of the tumor and the anal margin is ≤10cm;
4. ECOG score ≤2

(4) Imaging diagnostic analysis was cT1-3NxM0; (for Phase II/III) (5) CT examination of the chest and abdomen and pelvis showed no evidence of metastasis (6) Patients undergoing chemoradiotherapy and surgery

Exclusion Criteria:

1. History of malignant tumors in the past;
2. Diagnosis of simultaneous multiple primary colorectal cancer or other cancers;
3. History of chemotherapy or radiotherapy prior to this trial
4. Those with contraindications to laparoscopic surgery, such as severe cardiopulmonary insufficiency;
5. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc., requiring emergency surgery;
6. Pregnant or lactating women;
7. Evidence of distant metastases prior to surgery
8. T4b tumors were found to invade the uterus, vagina, bladder, seminal vesicles, prostate, bone, and pelvic plexus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with low- and medium-level rectal cancer treated with chemoradiotherapy and surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2024